CLINICAL TRIAL: NCT00967356
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Ascending Oral Doses of AZD5985 in Healthy Male Subjects
Brief Title: AZD5985 Single Ascending Dose Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated (halted prematurely) due to tolerability issues.
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, Christer Hultquist MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D2300C00002
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD5985
  Interventions: Drug: AZD5985
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5985 — Single dose-The starting dose will be 40 mg, oral suspension, with up to 8 dose escalations not exceeding AstraZeneca predefined upper exposure limits
  Arms: A
Drug: Placebo — Oral suspension
  Arms: B

SUMMARY:
The aims of this study are to assess the safety, tolerability and pharmacokinetics of single ascending oral doses of AZD5985 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedure
* Healthy male subjects aged 18 to 45 years (inclusive)
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder in the opinion of the investigator
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs or ECG at baseline in the opinion of the investigator
* Participation in another investigational drug study within 3 months before Visit 2 or participation in a methodological study (no drug) 1 month prior to Visit 2

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-08; Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Safety variables (ECG, adverse events, blood pressure, pulse, body temp, safety lab) | Frequent sampling occasions during study days

SECONDARY OUTCOMES:
Pharmacokinetic variables | Frequent sampling occasions during study days

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Marianne Hartford, Principal Investigator — AstraZeneca R&D, Mölndal, Sweden
Locations (1):
- Research Site, Gothenburg, Sweden